CLINICAL TRIAL: NCT03258710
Title: A Multi-centre, One-arm Prospective Study to Evaluate Efficacy and Safety of Switching From Entecavir (ETV) to Tenofovir Disoproxil Fumarate (TDF) in Japanese Chronic Hepatitis B HBeAg-positive and HBV-DNA Undetectable Subjects
Brief Title: A Study of Switching From Entecavir to Tenofovir Disoproxil Fumarate in Subjects With Chronic Hepatitis B
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 205883
Record Dates: First submitted 2017-08-21; First posted 2017-08-23 (Actual); Results first posted 2020-01-02 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Hepatitis B, Chronic
Keywords: Tenofovir Disoproxil Fumarate; safety; chronic hepatitis B; virological effect
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Tenofovir

STUDY DESIGN:
Intervention Model Description: This is a single arm study where on-going ETV treatment is switched to TDF treatment. There is no randomization in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All subjects treated with Tenofovir Disoproxil Fumarate (Experimental): Subjects with on-going ETV treatment will be switched to Tenofovir Disoproxil Fumarate treatment. Subjects will start TDF on the day ETV is discontinued, without having overlapping treatment periods. All subjects will receive one tablet of TDF 300 mg once daily orally for 96 weeks.
  Interventions: Drug: Tenofovir Disoproxil Fumarate

INTERVENTIONS:
Drug: Tenofovir Disoproxil Fumarate — Tenofovir Disoproxil Fumarate is a nucleos(t)ide analogue that inhibits HBV growth. All subjects will receive one tablet of TDF 300 mg once daily orally for 96 weeks.

SUMMARY:
Tenofovir Disoproxil Fumarate is a nucleos(t)ide analogue that inhibits Hepatitis B Virus (HBV) growth, and is marketed in Japan with an indication for inhibition of HBV growth in subjects with chronic hepatitis B associated with HBV growth and abnormal liver function. This study has been planned to evaluate the virological effects and safety of switching from ETV to TDF in chronic hepatitis B (hepatitis B e-antigen [HBeAg])-positive and HBV- deoxyribonucleic acid (DNA) undetectable subjects. This study is designed as a multi-center, one-arm, post-marketing clinical study to investigate the HBsAg reduction in subjects who have not achieved the long-term goal, the loss of hepatitis B surface antigen (HBsAg). The study will be conducted in HBeAg-positive and HBV-DNA undetectable subjects treated with ETV. After switching ETV to TDF, TDF will be administered for 96 weeks. Approximately 80 subjects will be screened to achieve 65 evaluable subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 20 to 69 years of age inclusive, at the time of signing the informed consent
* Male and female subjects. A female subject is eligible to participate if she is not pregnant and not breastfeeding, and at least one of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP), OR
  * A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 4 days after the last dose of study treatment
* Capable of giving signed informed consent form (ICF)
* Subjects with chronic hepatitis B (CHB) (excluding hospitalized subjects)
* Subjects treated with ETV for at least 2 years prior to initiation of study treatment.
* The serum HBV-DNA level at screening is below the limit of quantitation (< 2.1 Log10 copies/milliliter [mL] or < 20 international unit [IU]/mL).
* Subjects with serum HBeAg positive at screening
* Meet either of the following serum HBsAg levels at screening:

  * Serum HBsAg 80 < to < 800 IU/mL and fluctuation range is equal or more than -0.1 Log10 IU/mL per year
  * Serum HBsAg >=800 IU/mL
* Meet all of the following criteria at screening:

  * Creatinine clearance (CLcr) >=70 mL/minute. CLcr is calculated using the following Cockcroft-Gault formula.

Male: CLcr = (body weight in kilogram [kg] multiplied by [140 minus age in years]) divided by (72 multiplied by serum creatinine [milligram {mg}/deciliter {dL}]) Female: CLcr = CLcr (male) multiplied by 0.85

* Hemoglobin >= 8 gram/dL
* WBC >=1000 per cubic millimeter (mm^3)

Exclusion Criteria:

* QTc > 450 millisecond (msec) or > 480 msec for subjects with bundle branch block
* Received any interferon or Hepatitis B vaccine therapy within 24 weeks prior to initiation of the study treatment.
* Received overdose of nonsteroidal anti-inflammatory drugs (NSAIDs) (excluding temporary or topical use) within 7 days prior to initiation of the study treatment.
* Received any of the following drugs within 8 weeks prior to initiation of the study treatment (excluding topical products such as ointment and/or cream etc).

  * Drugs causing renal impairment (examples: aminoglycosides, amphotericin B, vancomycin, foscarnet, cisplatin, pentamidine, tacrolimus, cyclosporine, some contrast mediums [ionic high-osmolar contrast media, ionic low-osmolar contrast media]
  * Competitors of renal excretion (except temporary use, example: probenecid)
  * Immunosuppressants (examples: azathioprine, cycolphosphamide) or chemotherapeutics (example: etoposide)
  * Glucocorticoid preparation
* Received TDF, Adefovir pivoxil (ADV) or Tenofovir Alafenamide Fumarate (TAF) within 2 years prior to initiation of the study treatment
* Participation in another clinical study within 6 months prior to screening, or planned participation in another clinical study simultaneously with this study.
* Co-infection with human immunodeficiency virus (HIV) or hepatitis C virus (HCV)
* Subjects with serious complication other than compensated CHB (cancer, significant renal, cardiovascular, pulmonary, or neurological disease, uncontrollable diabetes, etc.)
* Received or have a plan for solid organ or bone marrow transplantation
* Has proximal tubulopathy.
* Subjects with decompensated CHB who meet the following: direct bilirubin > 1.5 times upper limit of normal (ULN), Prothrombin Time (PT) < 60%, platelets < 75,000/mm3 and serum albumin < 3.0 g/dL
* Autoimmune hepatitis (Antinuclear titer > 1:160), excluding CHB
* Subjects with or suspected of having hepatocellular carcinoma (HCC) (including both primary and metastatic) from diagnostic imaging at screening, or with serum alpha-fetoprotein (AFP) > 50 nanogram (ng)/mL at screening
* History of HCC (except subjects who underwent resection or received curative treatment by radiofrequency, and with AFP <=10 ng/mL at screening)
* Woman who is pregnant, possibly pregnant, lactating or planning a pregnancy during the study period.
* Psychiatry disorder or cognitive disorder that may affect the subject's ability to give informed consent or to follow specified study procedures.
* Subjects with a history of alcohol or drug abuse
* Subjects whom the investigator (or sub-investigator) considers ineligible for the study.
* Subjects with hypersensitivity to study treatments or their components, nucleoside and/or nucleotide analogues. Subjects with drug allergy that, in the investigator's (sub-investigator's) [or medical monitor's] opinion, labeled contraindication for participation in the study, or other allergy.

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2018-12-28 (Actual); Study Completion 2019-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- Japan (12):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Ehime
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Nagasaki
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Tottori

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Suzuki F, Suzuki Y, Karino Y, Tanaka Y, Kurosaki M, Yatsuhashi H, Atarashi T, Atsukawa M, Watanabe T, Enomoto M, Kudo M, Maeda N, Kohno H, Joko K, Michitaka K, Miki K, Takahashi K, Ide T, Fujiyama S, Kohno T, Itoh H, Tsukamoto S, Suzuki Y, Kawano Y, Sugiura W, Kumada H. Switching from entecavir to tenofovir disoproxil fumarate for HBeAg-positive chronic hepatitis B patients: a phase 4, prospective study. BMC Gastroenterol. 2021 Dec 20;21(1):489. doi: 10.1186/s12876-021-02008-9. PMID 34930140

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multi-center, single-arm study to assess efficacy and safety of tenofovir disoproxil fumarate (TDF) by switching at Day 1 from entecavir hydrate (ETV) to TDF in chronic hepatitis B envelope antigen (HBeAg)-positive and hepatitis B virus-deoxyribonucleic acid (HBV-DNA) undetectable participants.
Pre-assignment Details: A total of 75 participants were enrolled in the study.
Groups:
- Tenofovir Disoproxil Fumarate: Participants with on-going ETV treatment were switched to TDF treatment on Day 1. Participants then started with TDF on the day ETV was discontinued, without any overlapping treatment periods. All participants received one tablet of TDF 300 milligram (mg) once daily orally for 96 weeks.
Period: Overall Study
Arm/Group | Tenofovir Disoproxil Fumarate
Started | 75
Completed | 72
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Protocol-defined stopping criteria | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 75
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.4 (9.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 55
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian-East Asian Heritage | 4
  Asian-Japanese Heritage | 71

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved 0.25 Logarithm to the Base 10 (Log10) Hepatitis B Surface Antigen (HBsAg) Reduction From the Baseline at Week 48
Description: Blood samples were collected to evaluate the HBsAg reduction from Baseline at Week 48. HBsAg reduction potential was obtained by evaluating log10 observation values minus log10 Baseline values. The HBsAg responder values were<=-0.25 log10 and non-responder values were >-0.25 log10 . Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Full analysis set (FAS) Population is defined as population of all participants enrolled in the study, excluding those who meet either of the following criteria: who have not received any dose of study treatment and who have no efficacy data (HBsAg, HBV-DNA, hepatitis B core-related antigen [HBcrAg], HBeAg, hepatitis B surface antibody [HBsAb],Hepatitis B envelope antibody [HBeAb], alanine aminotransferase [ALT]) from at least 15 days after the start of study treatment. Data for HBsAg responders have been presented.
Time Frame: Baseline (Day 1, Pre-dose) and at Week 48
Population: FAS Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 74
Percentage of Participants
  <= -0.25 log10 | 4 [0.8 to 11.4]
  > -0.25 log10 | 96 [88.6 to 99.2]

2. Secondary Outcome: Percentage of Participants Who Achieved 0.25 Log10 HBsAg Reduction From the Baseline at Weeks 24 and 96
Description: Blood samples were collected to evaluate the HBsAg reduction potential from Baseline at Weeks 24 and 96. HBsAg reduction potential was obtained by evaluating log10 observation values minus log10 Baseline values. Data for HBsAg responders have been presented. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose) and at Weeks 24 and 96
Population: FAS Population.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 74
Percentage of Participants
  Week 24 | 1 [0.0 to 7.3]
  Week 96 | 12 [5.7 to 21.8]

3. Secondary Outcome: Percentage of Participants Who Achieved HBsAg Loss at Weeks 24, 48 and 96
Description: Blood samples were collected to evaluate the percentage of participants with HBsAg loss at Weeks 24, 48 and 96. A 'Loss' of HBsAg means antigen is negative. HBsAg loss percentage is defined as number of participants with HBsAg loss divided by number of participants with positive HBsAg at Baseline. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: At Weeks 24, 48 and 96
Population: FAS Population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 74
Percentage of Participants
  Week 24 | 0
  Week 48 | 0
  Week 96 | 0

4. Secondary Outcome: Percentage of Participants Who Achieved HBsAg/Ab Seroconversion at Weeks 24, 48 and 96
Description: Blood samples were collected to evaluate the percentage of participants who achieved HBsAg/Ab seroconversion at Weeks 24, 48 and 96. Seroconversion of HBsAg means antigen is negative and antibody is positive. HBsAg Seroconversion percentage is defined as number of participants with HBsAg/Ab Seroconversion divided by number of participants with positive HBsAg and Negative HBsAb at Baseline. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: At Weeks 24, 48 and 96
Population: FAS Population. Only those participants with data available at specified data points were analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 73
Percentage of Participants
  Week 24 | 0
  Week 48 | 0
  Week 96 | 0

5. Secondary Outcome: Percentage of Participants Who Achieved HBeAg Loss at Weeks 24, 48 and 96
Description: Blood samples were collected to evaluate the percentage of participants with HBeAg loss at Weeks 24, 48 and 96. A 'Loss' of HBeAg means antigen is negative. HBeAg Loss percentage is defined as number of participants with HBeAg loss divided by number of participants with positive HBeAg at Baseline. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: At Weeks 24, 48 and 96
Population: FAS Population. Only those participants with data available at specified data points were analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 69
Percentage of Participants
  Week 24 | 12
  Week 48 | 12
  Week 96 | 25

6. Secondary Outcome: Percentage of Participants Who Achieved HBeAg/Ab Seroconversion at Weeks 24, 48 and 96
Description: Blood samples were collected to evaluate the percentage of participants who achieved HBeAg/Ab seroconversion at Weeks 24, 48 and 96. Seroconversion of HBeAg means antigen is negative and antibody is positive. HBeAg Seroconversion percentage is defined as number of participants with HBeAg/Ab Seroconversion divided by number of participants with positive HBeAg and Negative HBeAb at Baseline. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: At Weeks 24, 48 and 96
Population: FAS Population. Only those participants with data available at specified data points were analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 53
Percentage of Participants
  Week 24 | 8
  Week 48 | 13
  Week 96 | 25

7. Secondary Outcome: Change From Baseline Log Values for HBsAg Titer at Weeks 24, 48 and 96
Description: Blood samples were collected to evaluate the HBsAg titer at Weeks 24, 48 and 96. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1, Pre-dose) and at Weeks 24, 48 and 96
Population: FAS Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: Log Kilo International Units per Liter
Arm/Group | Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 74
Log Kilo International Units per Liter
  Week 24, n=74 | -0.049 (0.0913)
  Week 48, n=73: number analyzed (Participants) | 73
  Week 48, n=73 | -0.114 (0.0837)
  Week 96, n=72: number analyzed (Participants) | 72
  Week 96, n=72 | -0.139 (0.1207)

8. Secondary Outcome: Change From Baseline Log Values for HBcrAg Titer at Weeks 24, 48 and 96
Description: Blood samples were collected to evaluate the HBcrAg titer at Weeks 24, 48 and 96. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1, Pre-dose) and at Weeks 24, 48 and 96
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Log Kilounits per Liter
Arm/Group | Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 74
Log Kilounits per Liter
  Week 24, n=74 | -0.12 (0.232)
  Week 48, n=73: number analyzed (Participants) | 73
  Week 48, n=73 | -0.17 (0.286)
  Week 96, n=72: number analyzed (Participants) | 72
  Week 96, n=72 | -0.30 (0.360)

9. Secondary Outcome: Number of Participants Who Reported Serious Adverse Events (SAEs) and Non-serious Adverse Events (Non-SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. A SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect, associated with liver injury and impaired liver function or any other situations as per medical or scientific judgement. Safety Population consists of participants who have received at least one dose of study treatment after enrolment.
Time Frame: Up to Week 96
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 75
Participants
  Any SAE | 2
  Any non-SAE | 36

10. Secondary Outcome: Absolute Values for Clinical Chemistry Parameter: Alpha-fetoprotein (AFP)
Description: Blood samples were collected for the analysis of clinical chemistry parameter, AFP. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose) and at Weeks 4, 12, 24, 36, 48, 60, 72, 84 and 96
Population: Safety Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: Micrograms per liter
Arm/Group | Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 75
Micrograms per liter
  Baseline (Day 1), n=75 | 3.13 (1.474)
  Week 4, n=75 | 3.39 (1.507)
  Week 12, n=74: number analyzed (Participants) | 74
  Week 12, n=74 | 3.46 (1.642)
  Week 24, n=74: number analyzed (Participants) | 74
  Week 24, n=74 | 3.50 (1.597)
  Week 36, n=73: number analyzed (Participants) | 73
  Week 36, n=73 | 3.48 (1.578)
  Week 48, n=73: number analyzed (Participants) | 73
  Week 48, n=73 | 3.55 (1.693)
  Week 60, n=73: number analyzed (Participants) | 73
  Week 60, n=73 | 3.50 (1.683)
  Week 72, n=73: number analyzed (Participants) | 73
  Week 72, n=73 | 3.27 (1.499)
  Week 84, n=72: number analyzed (Participants) | 72
  Week 84, n=72 | 3.10 (1.478)
  Week 96, n=72: number analyzed (Participants) | 72
  Week 96, n=72 | 3.18 (1.537)

11. Secondary Outcome: Absolute Values for Clinical Chemistry Parameters: Albumin and Total Protein
Description: Blood samples were collected for the analysis of clinical chemistry parameters: albumin and total protein. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose) and at Weeks 4, 12, 24, 36, 48, 60, 72, 84 and 96
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 75
Grams per liter
  Albumin, Baseline (Day 1), n=75 | 44.7 (2.60)
  Albumin, Week 4, n=75 | 44.9 (2.21)
  Albumin, Week 12, n=74: number analyzed (Participants) | 74
  Albumin, Week 12, n=74 | 45.2 (2.17)
  Albumin, Week 24, n=74: number analyzed (Participants) | 74
  Albumin, Week 24, n=74 | 44.5 (2.18)
  Albumin, Week 36, n=73: number analyzed (Participants) | 73
  Albumin, Week 36, n=73 | 44.2 (2.11)
  Albumin, Week 48, n=73: number analyzed (Participants) | 73
  Albumin, Week 48, n=73 | 44.8 (2.20)
  Albumin, Week 60, n=73: number analyzed (Participants) | 73
  Albumin, Week 60, n=73 | 45.1 (1.88)
  Albumin, Week 72, n=73: number analyzed (Participants) | 73
  Albumin, Week 72, n=73 | 44.9 (2.14)
  Albumin, Week 84, n=72: number analyzed (Participants) | 72
  Albumin, Week 84, n=72 | 44.6 (2.05)
  Albumin, Week 96, n=72: number analyzed (Participants) | 72
  Albumin, Week 96, n=72 | 45.4 (2.26)
  Total protein, Baseline (Day 1) n=75 | 72.4 (4.28)
  Total protein, Week 4, n=75 | 72.6 (3.81)
  Total protein, Week 12, n=74: number analyzed (Participants) | 74
  Total protein, Week 12, n=74 | 73.1 (3.93)
  Total protein, Week 24, n=74: number analyzed (Participants) | 74
  Total protein, Week 24, n=74 | 72.0 (3.86)
  Total protein, Week 36, n=73: number analyzed (Participants) | 73
  Total protein, Week 36, n=73 | 71.7 (3.76)
  Total protein, Week 48, n=73: number analyzed (Participants) | 73
  Total protein, Week 48, n=73 | 72.6 (4.12)
  Total protein, Week 60, n=73: number analyzed (Participants) | 73
  Total protein, Week 60, n=73 | 72.8 (4.08)
  Total protein, Week 72, n=73: number analyzed (Participants) | 73
  Total protein, Week 72, n=73 | 72.4 (4.32)
  Total protein, Week 84, n=72: number analyzed (Participants) | 72
  Total protein, Week 84, n=72 | 72.4 (4.35)
  Total protein, Week 96, n=72: number analyzed (Participants) | 72
  Total protein, Week 96, n=72 | 73.0 (4.07)

12. Secondary Outcome: Absolute Values for Clinical Chemistry Parameters: Alkaline Phosphate (ALP), Alanine Amino Transferase (ALT), Aspartate Amino Transferase (AST), Creatinine Kinase (CPK), Gamma Glutamyl Transferase (GGT) and Lactate Dehydrogenase (LDH)
Description: Blood samples were collected for the analysis of clinical chemistry parameters: ALP, ALT, AST, CPK, GGT and LDH. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose) and at Weeks 4, 12, 24, 36, 48, 60, 72, 84 and 96
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 75
International units per liter
  ALP, Baseline (Day 1), n=75 | 210.4 (62.87)
  ALP, Week 4, n=75 | 227.6 (70.27)
  ALP, Week 12, n=74: number analyzed (Participants) | 74
  ALP, Week 12, n=74 | 243.1 (76.26)
  ALP, Week 24, n=74: number analyzed (Participants) | 74
  ALP, Week 24, n=74 | 242.1 (77.76)
  ALP, Week 36, n=73: number analyzed (Participants) | 73
  ALP, Week 36, n=73 | 245.3 (75.15)
  ALP, Week 48, n=73: number analyzed (Participants) | 73
  ALP, Week 48, n=73 | 249.4 (73.17)
  ALP, Week 60, n=73: number analyzed (Participants) | 73
  ALP, Week 60, n=73 | 253.1 (75.62)
  ALP, Week 72, n=73: number analyzed (Participants) | 73
  ALP, Week 72, n=73 | 249.2 (72.56)
  ALP, Week 84, n=72: number analyzed (Participants) | 72
  ALP, Week 84, n=72 | 237.6 (69.60)
  ALP, Week 96, n=72: number analyzed (Participants) | 72
  ALP, Week 96, n=72 | 237.7 (72.92)
  ALT, Baseline (Day 1), n=75 | 23.5 (18.13)
  ALT, Week 4, n=75 | 28.3 (19.82)
  ALT, Week 12, n=74: number analyzed (Participants) | 74
  ALT, Week 12, n=74 | 27.9 (16.48)
  ALT, Week 24, n=74: number analyzed (Participants) | 74
  ALT, Week 24, n=74 | 27.5 (19.09)
  ALT, Week 36, n=73: number analyzed (Participants) | 73
  ALT, Week 36, n=73 | 25.9 (14.70)
  ALT, Week 48, n=73: number analyzed (Participants) | 73
  ALT, Week 48, n=73 | 27.0 (13.14)
  ALT, Week 60, n=73: number analyzed (Participants) | 73
  ALT, Week 60, n=73 | 26.6 (12.65)
  ALT, Week 72, n=73: number analyzed (Participants) | 73
  ALT, Week 72, n=73 | 24.2 (9.16)
  ALT, Week 84, n=72: number analyzed (Participants) | 72
  ALT, Week 84, n=72 | 26.3 (20.75)
  ALT, Week 96, n=72: number analyzed (Participants) | 72
  ALT, Week 96, n=72 | 26.4 (25.60)
  AST, Baseline (Day 1), n=75 | 22.7 (8.80)
  AST, Week 4, n=75 | 26.1 (8.70)
  AST, Week 12, n=74: number analyzed (Participants) | 74
  AST, Week 12, n=74 | 25.8 (8.34)
  AST, Week 24, n=74: number analyzed (Participants) | 74
  AST, Week 24, n=74 | 25.5 (9.31)
  AST, Week 36, n=73: number analyzed (Participants) | 73
  AST, Week 36, n=73 | 24.6 (7.88)
  AST, Week 48, n=73: number analyzed (Participants) | 73
  AST, Week 48, n=73 | 25.7 (7.58)
  AST, Week 60, n=73: number analyzed (Participants) | 73
  AST, Week 60, n=73 | 25.1 (6.23)
  AST, Week 72, n=73: number analyzed (Participants) | 73
  AST, Week 72, n=73 | 24.1 (5.25)
  AST, Week 84, n=72: number analyzed (Participants) | 72
  AST, Week 84, n=72 | 25.0 (10.38)
  AST, Week 96, n=72: number analyzed (Participants) | 72
  AST, Week 96, n=72 | 24.9 (12.03)
  CPK, Baseline (Day 1), n=75 | 138.9 (100.01)
  CPK, Week 4, n=75 | 151.0 (113.92)
  CPK, Week 12, n=74: number analyzed (Participants) | 74
  CPK, Week 12, n=74 | 144.5 (148.47)
  CPK, Week 24, n=74: number analyzed (Participants) | 74
  CPK, Week 24, n=74 | 127.9 (56.20)
  CPK, Week 36, n=73: number analyzed (Participants) | 73
  CPK, Week 36, n=73 | 131.9 (79.25)
  CPK, Week 48, n=73: number analyzed (Participants) | 73
  CPK, Week 48, n=73 | 148.7 (106.89)
  CKP, Week 60, n=73: number analyzed (Participants) | 73
  CKP, Week 60, n=73 | 134.1 (65.76)
  CKP, Week 72, n=73: number analyzed (Participants) | 73
  CKP, Week 72, n=73 | 143.3 (81.86)
  CKP, Week 84, n=72: number analyzed (Participants) | 72
  CKP, Week 84, n=72 | 127.4 (60.37)
  CKP, Week 96, n=72: number analyzed (Participants) | 72
  CKP, Week 96, n=72 | 132.3 (67.94)
  GGT, Baseline (Day 1), n=75 | 30.9 (24.23)
  GGT, Week 4, n=75 | 31.6 (27.23)
  GGT, Week 12, n=74: number analyzed (Participants) | 74
  GGT, Week 12, n=74 | 31.5 (31.14)
  GGT, Week 24, n=74: number analyzed (Participants) | 74
  GGT, Week 24, n=74 | 30.4 (28.57)
  GGT, Week 36, n=73: number analyzed (Participants) | 73
  GGT, Week 36, n=73 | 27.6 (24.30)
  GGT, Week 48, n=73: number analyzed (Participants) | 73
  GGT, Week 48, n=73 | 27.8 (22.60)
  GGT, Week 60, n=73: number analyzed (Participants) | 73
  GGT, Week 60, n=73 | 28.2 (24.67)
  GGT, Week 72, n=73: number analyzed (Participants) | 73
  GGT, Week 72, n=73 | 25.6 (16.94)
  GGT, Week 84, n=72: number analyzed (Participants) | 72
  GGT, Week 84, n=72 | 27.4 (25.22)
  GGT, Week 96, n=72: number analyzed (Participants) | 72
  GGT, Week 96, n=72 | 27.8 (23.75)
  LDH, Baseline (Day 1), n=75 | 165.2 (30.53)
  LDH, Week 4, n=75 | 173.9 (35.23)
  LDH, Week 12, n=74: number analyzed (Participants) | 74
  LDH, Week 12, n=74 | 171.0 (32.19)
  LDH, Week 24, n=74: number analyzed (Participants) | 74
  LDH, Week 24, n=74 | 169.4 (28.94)
  LDH, Week 36, n=73: number analyzed (Participants) | 73
  LDH, Week 36, n=73 | 170.3 (28.91)
  LDH, Week 48, n=73: number analyzed (Participants) | 73
  LDH, Week 48, n=73 | 175.3 (33.33)
  LDH, Week 60, n=73: number analyzed (Participants) | 73
  LDH, Week 60, n=73 | 174.4 (33.12)
  LDH, Week 72, n=73: number analyzed (Participants) | 73
  LDH, Week 72, n=73 | 174.6 (32.97)
  LDH, Week 84, n=72: number analyzed (Participants) | 72
  LDH, Week 84, n=72 | 172.7 (34.58)
  LDH, Week 96, n=72: number analyzed (Participants) | 72
  LDH, Week 96, n=72 | 173.2 (34.08)

13. Secondary Outcome: Absolute Values for Clinical Chemistry Parameters: Amylase and Lipase
Description: Blood samples were collected for the analysis of clinical chemistry parameters: amylase and lipase. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose) and at Weeks 4, 12, 24, 36, 48, 60, 72, 84 and 96
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 75
Units per liter
  Amylase, Baseline (Day 1), n=75 | 87.3 (26.00)
  Amylase, Week 4, n=75 | 89.5 (24.99)
  Amylase, Week 12, n=74: number analyzed (Participants) | 74
  Amylase, Week 12, n=74 | 88.2 (26.21)
  Amylase, Week 24, n=74: number analyzed (Participants) | 74
  Amylase, Week 24, n=74 | 83.7 (23.30)
  Amylase, Week 36, n=73: number analyzed (Participants) | 73
  Amylase, Week 36, n=73 | 82.3 (24.29)
  Amylase, Week 48, n=73: number analyzed (Participants) | 73
  Amylase, Week 48, n=73 | 84.9 (26.08)
  Amylase, Week 60, n=73: number analyzed (Participants) | 73
  Amylase, Week 60, n=73 | 92.2 (32.20)
  Amylase, Week 72, n=73: number analyzed (Participants) | 73
  Amylase, Week 72, n=73 | 88.8 (27.87)
  Amylase, Week 84, n=72: number analyzed (Participants) | 72
  Amylase, Week 84, n=72 | 84.4 (24.93)
  Amylase, Week 96, n=72: number analyzed (Participants) | 72
  Amylase, Week 96, n=72 | 86.7 (32.31)
  Lipase, Baseline (Day 1), n=75 | 40.0 (17.99)
  Lipase, Week 4, n=75 | 41.9 (14.27)
  Lipase, Week 12, n=74: number analyzed (Participants) | 74
  Lipase, Week 12, n=74 | 39.1 (13.97)
  Lipase, Week 24, n=74: number analyzed (Participants) | 74
  Lipase, Week 24, n=74 | 36.0 (9.95)
  Lipase, Week 36, n=73: number analyzed (Participants) | 73
  Lipase, Week 36, n=73 | 36.9 (12.64)
  Lipase, Week 48, n=73: number analyzed (Participants) | 73
  Lipase, Week 48, n=73 | 36.2 (12.91)
  Lipase, Week 60, n=73: number analyzed (Participants) | 73
  Lipase, Week 60, n=73 | 39.1 (13.07)
  Lipase, Week 72, n=73: number analyzed (Participants) | 73
  Lipase, Week 72, n=73 | 37.1 (13.72)
  Lipase, Week 84, n=72: number analyzed (Participants) | 72
  Lipase, Week 84, n=72 | 33.5 (11.55)
  Lipase, Week 96, n=72: number analyzed (Participants) | 72
  Lipase, Week 96, n=72 | 34.2 (16.73)

14. Secondary Outcome: Absolute Values for Clinical Chemistry Parameters: Direct Bilirubin, Total Bilirubin, Creatinine and Uric Acid
Description: Blood samples were collected for the analysis of clinical chemistry parameters: direct bilirubin, total bilirubin, creatinine and uric acid. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose) and at Weeks 4, 12, 24, 36, 48, 60, 72, 84 and 96
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 75
Micromoles per liter
  Direct bilirubin, Baseline (Day 1), n=75 | 3.899 (2.0574)
  Direct bilirubin, Week 4, n=75 | 3.944 (1.6386)
  Direct bilirubin, Week 12, n=74: number analyzed (Participants) | 74
  Direct bilirubin, Week 12, n=74 | 3.928 (1.5943)
  Direct bilirubin, Week 24, n=74: number analyzed (Participants) | 74
  Direct bilirubin, Week 24, n=74 | 4.021 (1.9493)
  Direct bilirubin, Week 36, n=73: number analyzed (Participants) | 73
  Direct bilirubin, Week 36, n=73 | 3.959 (1.9304)
  Direct bilirubin, Week 48, n=73: number analyzed (Participants) | 73
  Direct bilirubin, Week 48, n=73 | 4.029 (2.1015)
  Direct bilirubin, Week 60, n=73: number analyzed (Participants) | 73
  Direct bilirubin, Week 60, n=73 | 3.607 (1.4409)
  Direct bilirubin, Week 72, n=73: number analyzed (Participants) | 73
  Direct bilirubin, Week 72, n=73 | 3.959 (1.7540)
  Direct bilirubin, Week 84, n=72: number analyzed (Participants) | 72
  Direct bilirubin, Week 84, n=72 | 3.919 (1.7560)
  Direct bilirubin, Week 96, n=72: number analyzed (Participants) | 72
  Direct bilirubin, Week 96, n=72 | 4.418 (1.8765)
  Total bilirubin, Baseline (Day 1), n=75 | 10.693 (5.4663)
  Total bilirubin, Week 4, n=75 | 10.009 (4.1478)
  Total bilirubin, Week 12, n=74: number analyzed (Participants) | 74
  Total bilirubin, Week 12, n=74 | 9.890 (4.1528)
  Total bilirubin, Week 24, n=74: number analyzed (Participants) | 74
  Total bilirubin, Week 24, n=74 | 10.584 (5.4641)
  Total bilirubin, Week 36, n=73: number analyzed (Participants) | 73
  Total bilirubin, Week 36, n=73 | 10.518 (5.2834)
  Total bilirubin, Week 48, n=73: number analyzed (Participants) | 73
  Total bilirubin, Week 48, n=73 | 10.635 (5.6373)
  Total bilirubin, Week 60, n=73: number analyzed (Participants) | 73
  Total bilirubin, Week 60, n=73 | 9.557 (3.7684)
  Total bilirubin, Week 72, n=73: number analyzed (Participants) | 73
  Total bilirubin, Week 72, n=73 | 10.237 (5.0381)
  Total bilirubin, Week 84, n=72: number analyzed (Participants) | 72
  Total bilirubin, Week 84, n=72 | 10.284 (5.9340)
  Total bilirubin, Week 96, n=72: number analyzed (Participants) | 72
  Total bilirubin, Week 96, n=72 | 11.329 (4.4037)
  Creatinine, Baseline (Day 1), n=75 | 62.9997 (11.33874)
  Creatinine, Week 4, n=75 | 64.1666 (11.28624)
  Creatinine, Week 12, n=74: number analyzed (Participants) | 74
  Creatinine, Week 12, n=74 | 65.8102 (10.95564)
  Creatinine, Week 24, n=74: number analyzed (Participants) | 74
  Creatinine, Week 24, n=74 | 65.2965 (11.04922)
  Creatinine, Week 36, n=73: number analyzed (Participants) | 73
  Creatinine, Week 36, n=73 | 65.9852 (10.57867)
  Creatinine, Week 48, n=73: number analyzed (Participants) | 73
  Creatinine, Week 48, n=73 | 65.9125 (11.31592)
  Creatinine, Week 60, n=73: number analyzed (Participants) | 73
  Creatinine, Week 60, n=73 | 65.3191 (10.70634)
  Creatinine, Week 72, n=73: number analyzed (Participants) | 73
  Creatinine, Week 72, n=73 | 65.4887 (11.06350)
  Creatinine, Week 84, n=72: number analyzed (Participants) | 72
  Creatinine, Week 84, n=72 | 66.5578 (11.42181)
  Creatinine, Week 96, n=72: number analyzed (Participants) | 72
  Creatinine, Week 96, n=72 | 67.3436 (11.07035)
  Uric acid, Baseline (Day 1), n=75 | 333.0880 (71.24862)
  Uric acid, Week 4, n=75 | 322.9367 (67.10023)
  Uric acid, Week 12, n=74: number analyzed (Participants) | 74
  Uric acid, Week 12, n=74 | 323.3622 (73.51388)
  Uric acid, Week 24, n=74: number analyzed (Participants) | 74
  Uric acid, Week 24, n=74 | 321.3528 (70.76893)
  Uric acid, Week 36, n=73: number analyzed (Participants) | 73
  Uric acid, Week 36, n=73 | 320.9476 (70.10092)
  Uric acid, Week 48, n=73: number analyzed (Participants) | 73
  Uric acid, Week 48, n=73 | 320.8661 (67.21277)
  Uric acid, Week 60, n=73: number analyzed (Participants) | 73
  Uric acid, Week 60, n=73 | 309.3775 (62.83437)
  Uric acid, Week 72, n=73: number analyzed (Participants) | 73
  Uric acid, Week 72, n=73 | 318.0958 (71.99367)
  Uric acid, Week 84, n=72: number analyzed (Participants) | 72
  Uric acid, Week 84, n=72 | 318.0528 (66.72860)
  Uric acid, Week 96, n=72: number analyzed (Participants) | 72
  Uric acid, Week 96, n=72 | 328.0487 (71.10783)

15. Secondary Outcome: Absolute Values for Clinical Chemistry Parameters: Calcium, Chloride, Glucose, Potassium, Lactic Acid, Sodium, Phosphorus and Blood Urea Nitrogen (BUN)
Description: Blood samples were collected for the analysis of clinical chemistry parameters: calcium, chloride, glucose, potassium, lactic acid, sodium, phosphorus inorganic and BUN. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose) and at Weeks 4, 12, 24, 36, 48, 60, 72, 84 and 96
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 75
Millimoles per liter
  Calcium, Baseline (Day 1), n=75 | 2.290743 (0.0712447)
  Calcium, Week 4, n=75 | 2.272446 (0.0650823)
  Calcium, Week 12, n=74: number analyzed (Participants) | 74
  Calcium, Week 12, n=74 | 2.265393 (0.0642412)
  Calcium, Week 24, n=74: number analyzed (Participants) | 74
  Calcium, Week 24, n=74 | 2.251232 (0.0711166)
  Calcium, Week 36, n=73: number analyzed (Participants) | 73
  Calcium, Week 36, n=73 | 2.257121 (0.0674474)
  Calcium, Week 48, n=73: number analyzed (Participants) | 73
  Calcium, Week 48, n=73 | 2.297792 (0.0662944)
  Calcium, Week 60, n=73: number analyzed (Participants) | 73
  Calcium, Week 60, n=73 | 2.316932 (0.0668335)
  Calcium, Week 72, n=73: number analyzed (Participants) | 73
  Calcium, Week 72, n=73 | 2.297451 (0.0711492)
  Calcium, Week 84, n=72: number analyzed (Participants) | 72
  Calcium, Week 84, n=72 | 2.289856 (0.0621422)
  Calcium, Week 96, n=72: number analyzed (Participants) | 72
  Calcium, Week 96, n=72 | 2.306489 (0.0685384)
  Chloride, Baseline (Day 1), n=75 | 103.5 (2.09)
  Chloride, Week 4, n=75 | 103.3 (1.90)
  Chloride, Week 12, n=74: number analyzed (Participants) | 74
  Chloride, Week 12, n=74 | 103.5 (2.04)
  Chloride, Week 24, n=74: number analyzed (Participants) | 74
  Chloride, Week 24, n=74 | 103.9 (1.70)
  Chloride, Week 36, n=73: number analyzed (Participants) | 73
  Chloride, Week 36, n=73 | 104.0 (1.98)
  Chloride, Week 48, n=73: number analyzed (Participants) | 73
  Chloride, Week 48, n=73 | 103.6 (1.87)
  Chloride, Week 60, n=73: number analyzed (Participants) | 73
  Chloride, Week 60, n=73 | 103.6 (1.85)
  Chloride, Week 72, n=73: number analyzed (Participants) | 73
  Chloride, Week 72, n=73 | 104.1 (2.16)
  Chloride, Week 84, n=72: number analyzed (Participants) | 72
  Chloride, Week 84, n=72 | 104.9 (2.40)
  Chloride, Week 96, n=72: number analyzed (Participants) | 72
  Chloride, Week 96, n=72 | 104.3 (2.01)
  Glucose, Baseline (Day 1), n=75 | 5.832251 (1.3417805)
  Glucose, Week 4, n=75 | 5.704208 (1.0439295)
  Glucose, Week 12, n=74: number analyzed (Participants) | 74
  Glucose, Week 12, n=74 | 5.590757 (0.8796367)
  Glucose, Week 24, n=74: number analyzed (Participants) | 74
  Glucose, Week 24, n=74 | 5.652268 (0.9310549)
  Glucose, Week 36, n=73: number analyzed (Participants) | 73
  Glucose, Week 36, n=73 | 5.582937 (1.0191927)
  Glucose, Week 48, n=73: number analyzed (Participants) | 73
  Glucose, Week 48, n=73 | 5.709165 (0.8209347)
  Glucose, Week 60, n=73: number analyzed (Participants) | 73
  Glucose, Week 60, n=73 | 5.887862 (1.1524669)
  Glucose, Week 72, n=73: number analyzed (Participants) | 73
  Glucose, Week 72, n=73 | 5.801175 (0.9035958)
  Glucose, Week 84, n=72: number analyzed (Participants) | 72
  Glucose, Week 84, n=72 | 5.938799 (1.0721973)
  Glucose, Week 96, n=72: number analyzed (Participants) | 72
  Glucose, Week 96, n=72 | 5.544061 (0.6818280)
  Potassium, Baseline (Day 1), n=75 | 4.07 (0.258)
  Potassium, Week 4, n=75 | 4.07 (0.254)
  Potassium, Week 12, n=74: number analyzed (Participants) | 74
  Potassium, Week 12, n=74 | 4.04 (0.257)
  Potassium, Week 24, n=74: number analyzed (Participants) | 74
  Potassium, Week 24, n=74 | 4.03 (0.236)
  Potassium, Week 36, n=73: number analyzed (Participants) | 73
  Potassium, Week 36, n=73 | 4.02 (0.264)
  Potassium, Week 48, n=73: number analyzed (Participants) | 73
  Potassium, Week 48, n=73 | 4.05 (0.249)
  Potassium, Week 60, n=73: number analyzed (Participants) | 73
  Potassium, Week 60, n=73 | 4.09 (0.275)
  Potassium, Week 72, n=73: number analyzed (Participants) | 73
  Potassium, Week 72, n=73 | 4.10 (0.288)
  Potassium, Week 84, n=72: number analyzed (Participants) | 72
  Potassium, Week 84, n=72 | 4.03 (0.260)
  Potassium, Week 96, n=72: number analyzed (Participants) | 72
  Potassium, Week 96, n=72 | 4.05 (0.233)
  Lactic acid, Baseline (Day 1), n=75 | 1.10467 (0.397387)
  Lactic acid, Week 4, n=75 | 1.02342 (0.378255)
  Lactic acid, Week 12, n=74: number analyzed (Participants) | 74
  Lactic acid, Week 12, n=74 | 1.07535 (0.464637)
  Lactic acid, Week 24, n=74: number analyzed (Participants) | 74
  Lactic acid, Week 24, n=74 | 1.04970 (0.401795)
  Lactic acid, Week 36, n=73: number analyzed (Participants) | 73
  Lactic acid, Week 36, n=73 | 1.06089 (0.434265)
  Lactic acid, Week 48, n=73: number analyzed (Participants) | 73
  Lactic acid, Week 48, n=73 | 1.02865 (0.413619)
  Lactic acid, Week 60, n=73: number analyzed (Participants) | 73
  Lactic acid, Week 60, n=73 | 1.15182 (0.466672)
  Lactic acid, Week 72, n=73: number analyzed (Participants) | 73
  Lactic acid, Week 72, n=73 | 1.06332 (0.375955)
  Lactic acid, Week 84, n=72: number analyzed (Participants) | 72
  Lactic acid, Week 84, n=72 | 1.12526 (0.493101)
  Lactic acid, Week 96, n=72: number analyzed (Participants) | 72
  Lactic acid, Week 96, n=72 | 0.93703 (0.400024)
  Sodium, Baseline (Day 1), n=75 | 141.6 (1.64)
  Sodium, Week 4, n=75 | 141.9 (1.61)
  Sodium, Week 12, n=74: number analyzed (Participants) | 74
  Sodium, Week 12, n=74 | 142.3 (1.45)
  Sodium, Week 24, n=74: number analyzed (Participants) | 74
  Sodium, Week 24, n=74 | 142.2 (1.32)
  Sodium, Week 36, n=73: number analyzed (Participants) | 73
  Sodium, Week 36, n=73 | 142.0 (1.52)
  Sodium, Week 48, n=73: number analyzed (Participants) | 73
  Sodium, Week 48, n=73 | 142.0 (1.45)
  Sodium, Week 60, n=73: number analyzed (Participants) | 73
  Sodium, Week 60, n=73 | 142.2 (1.55)
  Sodium, Week 72, n=73: number analyzed (Participants) | 73
  Sodium, Week 72, n=73 | 142.0 (1.26)
  Sodium, Week 84, n=72: number analyzed (Participants) | 72
  Sodium, Week 84, n=72 | 142.0 (1.74)
  Sodium, Week 96, n=72: number analyzed (Participants) | 72
  Sodium, Week 96, n=72 | 141.3 (1.43)
  Phosphorus inorganic, Baseline (Day 1), n=75 | 1.072028 (0.1757407)
  Phosphorus inorganic, Week 4, n=75 | 1.031558 (0.1563869)
  Phosphorus inorganic, Week 12, n=74: number analyzed (Participants) | 74
  Phosphorus inorganic, Week 12, n=74 | 1.061206 (0.1621407)
  Phosphorus inorganic, Week 24, n=74: number analyzed (Participants) | 74
  Phosphorus inorganic, Week 24, n=74 | 1.052479 (0.1695973)
  Phosphorus inorganic, Week 36, n=73: number analyzed (Participants) | 73
  Phosphorus inorganic, Week 36, n=73 | 1.061589 (0.1529705)
  Phosphorus inorganic, Week 48, n=73: number analyzed (Participants) | 73
  Phosphorus inorganic, Week 48, n=73 | 1.073090 (0.1642529)
  Phosphorus inorganic, Week 60, n=73: number analyzed (Participants) | 73
  Phosphorus inorganic, Week 60, n=73 | 1.071320 (0.1738322)
  Phosphorus inorganic, Week 72, n=73: number analyzed (Participants) | 73
  Phosphorus inorganic, Week 72, n=73 | 1.082378 (0.1734792)
  Phosphorus inorganic, Week 84, n=72: number analyzed (Participants) | 72
  Phosphorus inorganic, Week 84, n=72 | 1.070952 (0.1739292)
  Phosphorus inorganic, Week 96, n=72: number analyzed (Participants) | 72
  Phosphorus inorganic, Week 96, n=72 | 1.095169 (0.1397279)
  BUN, Baseline (Day 1), n=75 | 4.89518 (1.278805)
  BUN, Week 4, n=75 | 4.80712 (1.270529)
  BUN, Week 12, n=74: number analyzed (Participants) | 74
  BUN, Week 12, n=74 | 4.86581 (1.389805)
  BUN, Week 24, n=74: number analyzed (Participants) | 74
  BUN, Week 24, n=74 | 4.96519 (1.315155)
  BUN, Week 36, n=73: number analyzed (Participants) | 73
  BUN, Week 36, n=73 | 4.86449 (1.433234)
  BUN, Week 48, n=73: number analyzed (Participants) | 73
  BUN, Week 48, n=73 | 4.71289 (1.240093)
  BUN, Week 60, n=73: number analyzed (Participants) | 73
  BUN, Week 60, n=73 | 4.84884 (1.312435)
  BUN, Week 72, n=73: number analyzed (Participants) | 73
  BUN, Week 72, n=73 | 4.86889 (1.090615)
  BUN, Week 84, n=72: number analyzed (Participants) | 72
  BUN, Week 84, n=72 | 4.70000 (1.441539)
  BUN, Week 96, n=72: number analyzed (Participants) | 72
  BUN, Week 96, n=72 | 4.65389 (1.214425)

16. Secondary Outcome: Absolute Values for Clinical Chemistry Parameter: Creatinine Clearance
Description: Blood samples were collected for the analysis of clinical chemistry parameter, creatinine clearance. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose) and at Weeks 4, 12, 24, 36, 48, 60, 72, 84 and 96
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Milliliters per minute
Arm/Group | Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 75
Milliliters per minute
  Baseline (Day 1), n=75 | 114.06 (23.849)
  Week 4, n=75 | 112.50 (25.283)
  Week 12, n=74: number analyzed (Participants) | 74
  Week 12, n=74 | 108.76 (24.634)
  Week 24, n=74: number analyzed (Participants) | 74
  Week 24, n=74 | 108.86 (24.963)
  Week 36, n=73: number analyzed (Participants) | 73
  Week 36, n=73 | 105.23 (23.739)
  Week 48, n=73: number analyzed (Participants) | 73
  Week 48, n=73 | 105.50 (24.333)
  Week 60, n=73: number analyzed (Participants) | 73
  Week 60, n=73 | 107.51 (25.719)
  Week 72, n=73: number analyzed (Participants) | 73
  Week 72, n=73 | 106.73 (24.278)
  Week 84, n=72: number analyzed (Participants) | 72
  Week 84, n=72 | 104.00 (23.511)
  Week 96, n=72: number analyzed (Participants) | 72
  Week 96, n=72 | 101.47 (23.705)

17. Secondary Outcome: Absolute Values for Clinical Chemistry Parameter: Glomerular Filtration Rate (GFR)
Description: Blood samples were collected for the analysis of clinical chemistry parameter, GFR. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose) and at Weeks 4, 12, 24, 36, 48, 60, 72, 84 and 96
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Milliliters per second per 1.73*meter^2
Arm/Group | Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 75
Milliliters per second per 1.73*meter^2
  Baseline (Day 1), n=75 | 1.46981 (0.260068)
  Week 4, n=75 | 1.43825 (0.260661)
  Week 12, n=74: number analyzed (Participants) | 74
  Week 12, n=74 | 1.39282 (0.241198)
  Week 24, n=74: number analyzed (Participants) | 74
  Week 24, n=74 | 1.40228 (0.238776)
  Week 36, n=73: number analyzed (Participants) | 73
  Week 36, n=73 | 1.37971 (0.235498)
  Week 48, n=73: number analyzed (Participants) | 73
  Week 48, n=73 | 1.38564 (0.250919)
  Week 60, n=73: number analyzed (Participants) | 73
  Week 60, n=73 | 1.39501 (0.246331)
  Week 72, n=73: number analyzed (Participants) | 73
  Week 72, n=73 | 1.38998 (0.243750)
  Week 84, n=72: number analyzed (Participants) | 72
  Week 84, n=72 | 1.36299 (0.233140)
  Week 96, n=72: number analyzed (Participants) | 72
  Week 96, n=72 | 1.34355 (0.239422)

18. Secondary Outcome: Percentage of Basophils at Indicated Time Points
Description: Blood samples were collected for the analysis of hematology parameter: basophils. Mean and standard deviation values for percentage of basophils reported was presented.
Time Frame: At Weeks 36, 48, 60, 72, 84 and 96
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Percentage of basophils
Arm/Group | Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 73
Percentage of basophils
  Week 36, n=32: number analyzed (Participants) | 32
  Week 36, n=32 | 0.46 (0.240)
  Week 48, n=73 | 0.49 (0.303)
  Week 60, n=73 | 0.57 (0.453)
  Week 72, n=73 | 0.50 (0.319)
  Week 84, n=72: number analyzed (Participants) | 72
  Week 84, n=72 | 0.54 (0.305)
  Week 96, n=72: number analyzed (Participants) | 72
  Week 96, n=72 | 0.57 (0.376)

19. Secondary Outcome: Percentage of Eosinophils at Indicated Time Points
Description: Blood samples were collected for the analysis of hematology parameter: eosinophils. Mean and standard deviation values for percentage of eosinophils reported was presented.
Time Frame: At Weeks 36 , 48, 60, 72, 84 and 96
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Percentage of eosinophils
Arm/Group | Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 73
Percentage of eosinophils
  Week 36, n=32: number analyzed (Participants) | 32
  Week 36, n=32 | 2.44 (1.767)
  Week 48, n=73 | 2.94 (2.667)
  Week 60, n=73 | 2.85 (2.298)
  Week 72, n=73 | 3.09 (2.519)
  Week 84, n=72: number analyzed (Participants) | 72
  Week 84, n=72 | 2.84 (2.042)
  Week 96, n=72: number analyzed (Participants) | 72
  Week 96, n=72 | 2.57 (2.145)

20. Secondary Outcome: Percentage of Lymphocytes at Indicated Time Points
Description: Blood samples were collected for the analysis of hematology parameter: lymphocytes. Mean and standard deviation values for percentage of lymphocytes reported was presented.
Time Frame: At Weeks 36, 48, 60, 72, 84 and 96
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Percentage of lymphocytes
Arm/Group | Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 73
Percentage of lymphocytes
  Week 36, n=32: number analyzed (Participants) | 32
  Week 36, n=32 | 33.34 (8.858)
  Week 48, n=73 | 32.39 (8.516)
  Week 60, n=73 | 32.73 (7.541)
  Week 72, n=73 | 32.29 (8.579)
  Week 84, n=72: number analyzed (Participants) | 72
  Week 84, n=72 | 31.94 (7.424)
  Week 96, n=72: number analyzed (Participants) | 72
  Week 96, n=72 | 32.98 (8.215)

21. Secondary Outcome: Percentage of Monocytes at Indicated Time Points
Description: Blood samples were collected for the analysis of hematology parameter: monocytes. Mean and standard deviation values for percentage of monocytes reported was presented.
Time Frame: At Weeks 36, 48, 60, 72, 84 and 96
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Percentage of monocytes
Arm/Group | Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 73
Percentage of monocytes
  Week 36, n=32: number analyzed (Participants) | 32
  Week 36, n=32 | 5.30 (1.492)
  Week 48, n=73 | 5.46 (1.598)
  Week 60, n=73 | 5.65 (1.430)
  Week 72, n=73 | 5.67 (1.814)
  Week 84, n=72: number analyzed (Participants) | 72
  Week 84, n=72 | 5.71 (1.562)
  Week 96, n=72: number analyzed (Participants) | 72
  Week 96, n=72 | 5.45 (1.475)

22. Secondary Outcome: Percentage of Total Neutrophils at Indicated Time Points
Description: Blood samples were collected for the analysis of hematology parameter: total neutrophils. Mean and standard deviation values for percentage of neutrophils reported was presented.
Time Frame: At Weeks 36, 48, 60, 72, 84 and 96
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Percentage of neutrophils
Arm/Group | Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 73
Percentage of neutrophils
  Week 36, n=32: number analyzed (Participants) | 32
  Week 36, n=32 | 58.46 (8.658)
  Week 48, n=73 | 58.72 (8.709)
  Week 60, n=73 | 58.20 (8.176)
  Week 72, n=73 | 58.45 (9.109)
  Week 84, n=72: number analyzed (Participants) | 72
  Week 84, n=72 | 58.97 (7.881)
  Week 96, n=72: number analyzed (Participants) | 72
  Week 96, n=72 | 58.43 (8.973)

23. Secondary Outcome: Absolute Values for Hematology Parameter: Hemoglobin
Description: Blood samples were collected for the analysis of hematology parameter, hemoglobin. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose) and at Weeks 4, 12, 24, 36, 48, 60, 72, 84 and 96
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 75
Grams per liter
  Baseline (Day 1), n=75 | 148.2 (13.13)
  Week 4, n=75 | 148.9 (13.40)
  Week 12, n=74: number analyzed (Participants) | 74
  Week 12, n=74 | 148.4 (14.41)
  Week 24, n=74: number analyzed (Participants) | 74
  Week 24, n=74 | 146.3 (14.28)
  Week 36, n=73: number analyzed (Participants) | 73
  Week 36, n=73 | 144.1 (15.58)
  Week 48, n=73: number analyzed (Participants) | 73
  Week 48, n=73 | 146.5 (15.81)
  Week 60, n=73: number analyzed (Participants) | 73
  Week 60, n=73 | 147.1 (14.93)
  Week 72, n=73: number analyzed (Participants) | 73
  Week 72, n=73 | 146.4 (14.95)
  Week 84, n=72: number analyzed (Participants) | 72
  Week 84, n=72 | 144.6 (16.01)
  Week 96, n=72: number analyzed (Participants) | 72
  Week 96, n=72 | 146.4 (16.07)

24. Secondary Outcome: Absolute Values for Hematology Parameter: Hematocrit
Description: Blood samples were collected for the analysis of hematology parameter, hematocrit. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose) and at Weeks 4, 12, 24, 36, 48, 60, 72, 84 and 96
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 75
Proportion of red blood cells in blood
  Baseline (Day 1), n=75 | 0.4393 (0.03331)
  Week 4, n=75 | 0.4441 (0.03475)
  Week 12, n=74: number analyzed (Participants) | 74
  Week 12, n=74 | 0.4452 (0.03679)
  Week 24, n=74: number analyzed (Participants) | 74
  Week 24, n=74 | 0.4367 (0.03550)
  Week 36, n=73: number analyzed (Participants) | 73
  Week 36, n=73 | 0.4283 (0.04156)
  Week 48, n=73: number analyzed (Participants) | 73
  Week 48, n=73 | 0.4350 (0.03942)
  Week 60, n=73: number analyzed (Participants) | 73
  Week 60, n=73 | 0.4398 (0.03940)
  Week 72, n=73: number analyzed (Participants) | 73
  Week 72, n=73 | 0.4391 (0.03817)
  Week 84, n=72: number analyzed (Participants) | 72
  Week 84, n=72 | 0.4339 (0.04070)
  Week 96, n=72: number analyzed (Participants) | 72
  Week 96, n=72 | 0.4355 (0.04159)

25. Secondary Outcome: Absolute Values for Hematology Parameters: Platelet Count and White Blood Cell (WBC) Count
Description: Blood samples were collected for the analysis of hematology parameters: platelet count and WBC count. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose) and at Weeks 4, 12, 24, 36, 48, 60, 72, 84 and 96
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Giga cells per liter
Arm/Group | Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 75
Giga cells per liter
  Platelet count, Baseline (Day 1), n=75 | 226.7 (53.40)
  Platelet count, Week 4, n=75 | 227.1 (57.44)
  Platelet count, Week 12, n=74: number analyzed (Participants) | 74
  Platelet count, Week 12, n=74 | 228.9 (57.67)
  Platelet count, Week 24, n=74: number analyzed (Participants) | 74
  Platelet count, Week 24, n=74 | 226.1 (55.46)
  Platelet count, Week 36, n=73: number analyzed (Participants) | 73
  Platelet count, Week 36, n=73 | 231.4 (65.32)
  Platelet count, Week 48, n=73: number analyzed (Participants) | 73
  Platelet count, Week 48, n=73 | 229.9 (57.37)
  Platelet count, Week 60, n=73: number analyzed (Participants) | 73
  Platelet count, Week 60, n=73 | 231.8 (56.11)
  Platelet count, Week 72, n=73: number analyzed (Participants) | 73
  Platelet count, Week 72, n=73 | 224.9 (53.00)
  Platelet count, Week 84, n=72: number analyzed (Participants) | 72
  Platelet count, Week 84, n=72 | 224.8 (57.64)
  Platelet count, Week 96, n=72: number analyzed (Participants) | 72
  Platelet count, Week 96, n=72 | 226.6 (54.72)
  WBC count, Baseline (Day 1), n=75 | 5.18 (1.558)
  WBC count, Week 4, n=75 | 5.21 (1.525)
  WBC count, Week 12, n=74: number analyzed (Participants) | 74
  WBC count, Week 12, n=74 | 5.30 (1.380)
  WBC count, Week 24, n=74: number analyzed (Participants) | 74
  WBC count, Week 24, n=74 | 5.06 (1.279)
  WBC count, Week 36, n=73: number analyzed (Participants) | 73
  WBC count, Week 36, n=73 | 4.99 (1.320)
  WBC count, Week 48, n=73: number analyzed (Participants) | 73
  WBC count, Week 48, n=73 | 5.16 (1.674)
  WBC count, Week 60, n=73: number analyzed (Participants) | 73
  WBC count, Week 60, n=73 | 4.84 (1.247)
  WBC count, Week 72, n=73: number analyzed (Participants) | 73
  WBC count, Week 72, n=73 | 5.00 (1.372)
  WBC count, Week 84, n=72: number analyzed (Participants) | 72
  WBC count, Week 84, n=72 | 5.00 (1.338)
  WBC count, Week 96, n=72: number analyzed (Participants) | 72
  WBC count, Week 96, n=72 | 5.08 (1.583)

26. Secondary Outcome: Absolute Values for Hematology Parameter: Prothrombin Time
Description: Blood samples were collected for the analysis of hematology parameter, prothrombin time. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose) and at Weeks 4, 12, 24, 36, 48, 60, 72, 84 and 96
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 75
Seconds
  Baseline (Day 1), n=75 | 11.82 (0.632)
  Week 4, n=75 | 11.91 (0.679)
  Week 12, n=74: number analyzed (Participants) | 74
  Week 12, n=74 | 11.95 (0.642)
  Week 24, n=74: number analyzed (Participants) | 74
  Week 24, n=74 | 11.76 (0.627)
  Week 36, n=73: number analyzed (Participants) | 73
  Week 36, n=73 | 11.94 (0.720)
  Week 48, n=73: number analyzed (Participants) | 73
  Week 48, n=73 | 12.71 (0.681)
  Week 60, n=73: number analyzed (Participants) | 73
  Week 60, n=73 | 12.32 (0.613)
  Week 72, n=73: number analyzed (Participants) | 73
  Week 72, n=73 | 12.40 (0.615)
  Week 84, n=72: number analyzed (Participants) | 72
  Week 84, n=72 | 12.58 (0.684)
  Week 96, n=72: number analyzed (Participants) | 72
  Week 96, n=72 | 12.78 (0.766)

27. Secondary Outcome: Absolute Values for Hematology Parameter: Red Blood Cell (RBC) Count
Description: Blood samples were collected for the analysis of hematology parameter, RBC count. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose) and at Weeks 4, 12, 24, 36, 48, 60, 72, 84 and 96
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Trillion cells per liter
Arm/Group | Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 75
Trillion cells per liter
  Baseline (Day 1), n=75 | 4.785 (0.4087)
  Week 4, n=75 | 4.841 (0.4154)
  Week 12, n=74: number analyzed (Participants) | 74
  Week 12, n=74 | 4.865 (0.4358)
  Week 24, n=74: number analyzed (Participants) | 74
  Week 24, n=74 | 4.820 (0.4061)
  Week 36, n=73: number analyzed (Participants) | 73
  Week 36, n=73 | 4.704 (0.4473)
  Week 48, n=73: number analyzed (Participants) | 73
  Week 48, n=73 | 4.780 (0.4026)
  Week 60, n=73: number analyzed (Participants) | 73
  Week 60, n=73 | 4.819 (0.4288)
  Week 72, n=73: number analyzed (Participants) | 73
  Week 72, n=73 | 4.793 (0.4058)
  Week 84, n=72: number analyzed (Participants) | 72
  Week 84, n=72 | 4.757 (0.4314)
  Week 96, n=72: number analyzed (Participants) | 72
  Week 96, n=72 | 4.777 (0.4440)

28. Secondary Outcome: Number of Participants With Abnormal Urinalysis Values at Weeks 4, 12, 24, 36 and 48
Description: Urine samples were collected for analysis of urinalysis data for glucose, protein and urinary sediment by dipstick method. The urine sediments analyzed were amorphous phosphate crystals, amorphous urate crystals, bacteria, calcium oxalate crystals, ammonium magnesium phosphate, renal tubular epithelial cells (RTEC), fungi, hyaline casts, mucous threads, RBCs, spermatozoa, squamous epithelial cells (SEC), transitional epithelial cells (TEC), uric acid crystals (UAC) and WBCs. The dipstick test gives results in a semi-quantitative manner, and results for urinalysis parameters can be read as Trace, 1+, 2+ and 3+, indicating proportional concentrations in the urine sample. Results for RTEC, hyaline casts, RBC, SEC, TEC and WBC can be read as counts per field (some/ every/ whole field). Only abnormal parameters and participants with abnormal data has been reported.
Time Frame: Weeks 4, 12, 24, 36 and 48
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 75
Participants
  Amorphous phosphate crystals, Week 4, 1+ | 2
  Amorphous phosphate crystals, Week 12, 1+ | 2
  Amorphous phosphate crystals, Week 24, 1+ | 3
  Amorphous phosphate crystals, Week 36, 1+ | 2
  Amorphous phosphate crystals, Week 48, 1+ | 2
  Amorphous urate crystals, Week 4, 1+ | 3
  Amorphous urate crystals, Week 12, 1+ | 6
  Amorphous urate crystals, Week 24, 1+ | 8
  Amorphous urate crystals, Week 36, 1+ | 5
  Amorphous urate crystals, Week 48, 1+ | 5
  Bacteria, Week 4, 1+ | 5
  Bacteria, Week 12, 1+ | 11
  Bacteria, Week 24, 1+ | 6
  Bacteria, Week 24, 2+ | 2
  Bacteria, Week 36, 1+ | 8
  Bacteria, Week 48, 1+ | 11
  Bacteria, Week 48, 2+ | 1
  Calcium oxalate crystals, Week 4, 1+ | 11
  Calcium oxalate crystals, Week 12, 1+ | 9
  Calcium oxalate crystals, Week 24, 1+ | 14
  Calcium oxalate crystals, Week 36, 1+ | 15
  Calcium oxalate crystals, Week 48, 1+ | 10
  RTEC, Week 4, 0-0.1/Some Field | 23
  RTEC, Week 4, 0.2-0.4/Some Field | 5
  RTEC, Week 4, 1-2/Every Field | 1
  RTEC, Week 12, 0-0.1/Some Field | 25
  RTEC, Week 12, 0.2-0.4/Some Field | 4
  RTEC, Week 24, 0-0.1/Some Field | 19
  RTEC, Week 24, 0.2-0.4/Some Field | 2
  RTEC, Week 24, 1-2/Every Field | 1
  RTEC, Week 36, 0-0.1/Some Field | 19
  RTEC, Week 36, 0.2-0.4/Some Field | 2
  RTEC, Week 36, 1-2/Every Field | 1
  RTEC, Week 48, 0-0.1/Some Field | 21
  RTEC, Week 48, 0.2-0.4/Some Field | 5
  RTEC, Week 48, 1-2/Every Field | 3
  Fungi, Week 4, 1+ | 0
  Fungi, Week 12, 1+ | 0
  Fungi, Week 24, 1+ | 1
  Fungi, Week 36, 1+ | 0
  Fungi, Week 48, 1+ | 0
  Urine glucose, Week 4, 1+ | 1
  Urine glucose, Week 4, Trace | 1
  Urine glucose, Week 12, 2+ | 1
  Urine glucose, Week 12, Trace | 1
  Urine glucose, Week 24, 3+ | 1
  Urine glucose, Week 36, Trace | 2
  Urine glucose, Week 48, 1+ | 1
  Urine glucose, Week 48, 3+ | 1
  Urine glucose, Week 48, Trace | 1
  Hyaline casts, Week 4, 0-0.1/Some Field | 6
  Hyaline casts, Week 12, 0-0.1/Some Field | 3
  Hyaline casts, Week 12, 3-5/Whole Field | 2
  Hyaline casts, Week 24, 0-0.1/Some Field | 1
  Hyaline casts, Week 24, 1-2/Whole Field | 3
  Hyaline casts, Week 24, 3-5/Whole Field | 1
  Hyaline casts, Week 36, 0-0.1/Some Field | 1
  Hyaline casts, Week 36, 0.2-0.4/Some Field | 1
  Hyaline casts, Week 36, 1-2/Every Field | 1
  Hyaline casts, Week 36, 1-2/Whole Field | 1
  Hyaline casts, Week 48, 0-0.1/Some Field | 3
  Hyaline casts, Week 48, 0.2-0.4/Some Field | 1
  Mucus threads, Week 4, 1+ | 17
  Mucus threads, Week 12, 1+ | 21
  Mucus threads, Week 24, 1+ | 23
  Mucus threads, Week 36, 1+ | 25
  Mucus threads, Week 48, 1+ | 22
  Urine protein, Week 4, 1+ | 1
  Urine protein, Week 4, 2+ | 1
  Urine protein, Week 4, Trace | 15
  Urine protein, Week 12, 1+ | 2
  Urine protein, Week 12, Trace | 24
  Urine protein, Week 24, 1+ | 4
  Urine protein, Week 24, 2+ | 1
  Urine protein, Week 24, Trace | 28
  Urine protein, Week 36, 1+ | 3
  Urine protein, Week 36, 2+ | 1
  Urine protein, Week 36, Trace | 27
  Urine protein, Week 48, Trace | 15
  RBC, Week 4, 0-0.1/Some Field | 35
  RBC, Week 4, 0.2-0.4/Some Field | 20
  RBC, Week 4, 1-2/Every Field | 13
  RBC, Week 4, 3-5/Every Field | 4
  RBC, Week 4, 6-10/Every Field | 3
  RBC, Week 12, numerous/Every Field | 1
  RBC, Week 12, 0-0.1/Some Field | 33
  RBC, Week 12, 0.2-0.4/Some Field | 23
  RBC, Week 12, 1-2/Every Field | 11
  RBC, Week 12, 3-5/Every Field | 4
  RBC, Week 12, 6-10/Every Field | 1
  RBC, Week 12, 10-20/Every Field | 1
  RBC, Week 24, 0-0.1/Some Field | 40
  RBC, Week 24, 0.2-0.4/Some Field | 14
  RBC, Week 24, 1-2/Every Field | 14
  RBC, Week 24, 3-5/Every Field | 1
  RBC, Week 24, 6-10/Every Field | 2
  RBC, Week 24, 10-20/Every Field | 1
  RBC, Week 24, 20-30/Every Field | 2
  RBC, Week 36, 0-0.1/Some Field | 42
  RBC, Week 36, 0.2-0.4/Some Field | 20
  RBC, Week 36, 1-2/Every Field | 7
  RBC, Week 36, 3-5/Every Field | 1
  RBC, Week 36, 6-10/Every Field | 2
  RBC, Week 36, 10-20/Every Field | 1
  RBC, Week 48, 0-0.1/Some Field | 39
  RBC, Week 48, 0.2-0.4/Some Field | 14
  RBC, Week 48, 1-2/Every Field | 14
  RBC, Week 48, 3-5/Every Field | 3
  RBC, Week 48, 6-10/Every Field | 2
  RBC, Week 48, 10-20/Every Field | 1
  Spermatozoa, Week 4, 1+ | 1
  Spermatozoa, Week 12, 1+ | 0
  Spermatozoa, Week 24, 1+ | 2
  Spermatozoa, Week 36, 1+ | 3
  Spermatozoa, Week 48, 1+ | 0
  SEC, Week 4, 0-0.1/Some Field | 58
  SEC, Week 4, 0.2-0.4/Some Field | 7
  SEC, Week 4, 1-2/Every Field | 7
  SEC, Week 4, 3-5/Every Field | 2
  SEC, Week 4, 10-20/Every Field | 1
  SEC, Week 12, 0-0.1/Some Field | 54
  SEC, Week 12, 0.2-0.4/Some Field | 9
  SEC, Week 12, 1-2/Every Field | 6
  SEC, Week 12, 3-5/Every Field | 2
  SEC, Week 12, 6-10/Every Field | 1
  SEC, Week 12, 10-20/Every Field | 1
  SEC, Week 12, 30-50/Every Field | 1
  SEC, Week 24, 0-0.1/Some Field | 55
  SEC, Week 24, 0.2-0.4/Some Field | 6
  SEC, Week 24, 1-2/Every Field | 8
  SEC, Week 24, 3-5/Every Field | 1
  SEC, Week 24, 6-10/Every Field | 1
  SEC, Week 24, 10-20/Every Field | 2
  SEC, Week 24, 20-30/Every Field | 1
  SEC, Week 36, 0-0.1/Some Field | 59
  SEC, Week 36, 0.2-0.4/Some Field | 4
  SEC, Week 36, 1-2/Every Field | 9
  SEC, Week 36, 3-5/Every Field | 1
  SEC, Week 48, 0-0.1/Some Field | 58
  SEC, Week 48, 0.2-0.4/Some Field | 4
  SEC, Week 48, 1-2/Every Field | 5
  SEC, Week 48, 3-5/Every Field | 5
  SEC, Week 48, 6-10/Every Field | 1
  TEC, Week 4, 0-0.1/Some Field | 4
  TEC, Week 12, 0-0.1/Some Field | 4
  TEC, Week 24, 0-0.1/Some Field | 5
  TEC, Week 24, 0.2-0.4/Some Field | 2
  TEC, Week 36, 0-0.1/Some Field | 3
  TEC, Week 36, 0.2-0.4/Some Field | 1
  TEC, Week 36, 1-2/Every Field | 1
  TEC, Week 48, 0-0.1/Some Field | 5
  UAC, Week 4, 1+ | 0
  UAC, Week 12, 1+ | 0
  UAC, Week 24, 1+ | 0
  UAC, Week 36, 1+ | 2
  UAC, Week 48, 1+ | 1
  WBC, Week 4, 0-0.1/Some Field | 35
  WBC, Week 4, 0.2-0.4/Some Field | 27
  WBC, Week 4, 1-2/Every Field | 10
  WBC, Week 4, 3-5/Every Field | 1
  WBC, Week 4, 10-20/Every Field | 2
  WBC, Week 12, 0-0.1/Some Field | 37
  WBC, Week 12, 0.2-0.4/Some Field | 22
  WBC, Week 12, 1-2/Every Field | 8
  WBC, Week 12, 3-5/Every Field | 6
  WBC, Week 12, 6-10/Every Field | 1
  WBC, Week 24, 0-0.1/Some Field | 42
  WBC, Week 24, 0.2-0.4/Some Field | 20
  WBC, Week 24, 1-2/Every Field | 5
  WBC, Week 24, 3-5/Every Field | 3
  WBC, Week 24, 6-10/Every Field | 1
  WBC, Week 24, 10-20/Every Field | 2
  WBC, Week 24, 30-50/Every Field | 1
  WBC, Week 36, 0-0.1/Some Field | 45
  WBC, Week 36, 0.2-0.4/Some Field | 20
  WBC, Week 36, 1-2/Every Field | 1
  WBC, Week 36, 3-5/Every Field | 4
  WBC, Week 36, 6-10/Every Field | 2
  WBC, Week 36, 30-50/Every Field | 1
  WBC, Week 48, 0-0.1/Some Field | 43
  WBC, Week 48, 0.2-0.4/Some Field | 14
  WBC, Week 48, 1-2/Every Field | 11
  WBC, Week 48, 3-5/Every Field | 2
  WBC, Week 48, 6-10/Every Field | 2

29. Secondary Outcome: Number of Participants With Abnormal Urinalysis Values at Weeks 60, 72, 84 and 96
Description: as for outcome 28
Time Frame: Weeks 60, 72, 84 and 96
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 75
Participants
  Amorphous phosphate crystals, Week 60, 1+ | 2
  Amorphous phosphate crystals, Week 72, 1+ | 2
  Amorphous phosphate crystals, Week 84, 1+ | 2
  Amorphous urate crystals, Week 60, 1+ | 3
  Amorphous urate crystals, Week 72, 1+ | 2
  Amorphous urate crystals, Week 84, 1+ | 8
  Amorphous urate crystals, Week 96, 1+ | 3
  Bacteria, Week 60, 1+ | 15
  Bacteria, Week 72, 1+ | 7
  Bacteria, Week 72, 2+ | 3
  Bacteria, Week 84, 1+ | 9
  Bacteria, Week 84, 2+ | 2
  Bacteria, Week 96, 1+ | 9
  Bacteria, Week 96, 2+ | 1
  Calcium oxalate crystals, Week 60, 1+ | 14
  Calcium oxalate crystals, Week 72, 1+ | 12
  Calcium oxalate crystals, Week 84, 1+ | 16
  Calcium oxalate crystals, Week 96, 1+ | 4
  RTEC, Week 60, 0-0.1/Some Field | 19
  RTEC, Week 60, 0.2-0.4/Some Field | 7
  RTEC, Week 60, 1-2/Every Field | 1
  RTEC, Week 72, 0-0.1/Some Field | 14
  RTEC, Week 72, 0.2-0.4/Some Field | 5
  RTEC, Week 84, 0-0.1/Some Field | 9
  RTEC, Week 84, 0.2-0.4/Some Field | 4
  RTEC, Week 84, 1-2/Every Field | 2
  RTEC, Week 84, 3-5/Every Field | 1
  RTEC, Week 96, 0-0.1/Some Field | 15
  RTEC, Week 96, 0.2-0.4/Some Field | 2
  RTEC, Week 96, 1-2/Every Field | 1
  Urine glucose, Week 60, 3+ | 1
  Urine glucose, Week 72, 1+ | 1
  Urine glucose, Week 72, 2+ | 1
  Hyaline casts, Week 60, 0-0.1/Some Field | 4
  Hyaline casts, Week 72, 0-0.1/Some Field | 4
  Hyaline casts, Week 72, 0.2-0.4/Some Field | 1
  Hyaline casts, Week 84, 0-0.1/Some Field | 2
  Hyaline casts, Week 84, 1-2/Whole Field | 1
  Hyaline casts, Week 84, 3-5/Whole Field | 1
  Hyaline casts, Week 96, 0-0.1/Some Field | 2
  Hyaline casts, Week 96, 0.2-0.4/Some Field | 1
  Hyaline casts, Week 96, 3-5/Whole Field | 3
  Mucus threads, Week 60, 1+ | 27
  Mucus threads, Week 72, 1+ | 15
  Mucus threads, Week 84, 1+ | 18
  Mucus threads, Week 96, 1+ | 19
  Urine protein, Week 60, 1+ | 1
  Urine protein, Week 60, Trace | 11
  Urine protein, Week 72, 1+ | 2
  Urine protein, Week 72, Trace | 14
  Urine protein, Week 84, 1+ | 2
  Urine protein, Week 84, Trace | 17
  Urine protein, Week 96, 1+ | 3
  Urine protein, Week 96, Trace | 11
  RBC, Week 60, 0-0.1/Some Field | 35
  RBC, Week 60, 0.2-0.4/Some Field | 17
  RBC, Week 60, 1-2/Every Field | 12
  RBC, Week 60, 3-5/Every Field | 5
  RBC, Week 60, 6-10/Every Field | 1
  RBC, Week 60, 10-20/Every Field | 2
  RBC, Week 60, 30-50/Every Field | 1
  RBC, Week 72, 0-0.1/Some Field | 45
  RBC, Week 72, 0.2-0.4/Some Field | 11
  RBC, Week 72, 1-2/Every Field | 12
  RBC, Week 72, 3-5/Every Field | 3
  RBC, Week 72, 30-50/Every Field | 2
  RBC, Week 84, many/Every Field | 1
  RBC, Week 84, 0-0.1/Some Field | 40
  RBC, Week 84, 0.2-0.4/Some Field | 9
  RBC, Week 84, 1-2/Every Field | 15
  RBC, Week 84, 3-5/Every Field | 3
  RBC, Week 84, 6-10/Every Field | 2
  RBC, Week 84, 20-30/Every Field | 1
  RBC, Week 84, 30-50/Every Field | 1
  RBC, Week 96, many/Every Field | 1
  RBC, Week 96, 0-0.1/Some Field | 44
  RBC, Week 96, 0.2-0.4/Some Field | 11
  RBC, Week 96, 1-2/Every Field | 11
  RBC, Week 96, 3-5/Every Field | 4
  RBC, Week 96, 10-20/Every Field | 1
  Spermatozoa, Week 84, 1+ | 1
  SEC, Week 60, 0-0.1/Some Field | 52
  SEC, Week 60, 0.2-0.4/Some Field | 7
  SEC, Week 60, 1-2/Every Field | 9
  SEC, Week 60, 3-5/Every Field | 2
  SEC, Week 60, 10-20/Every Field | 2
  SEC, Week 60, 20-30/Every Field | 1
  SEC, Week 72, 0-0.1/Some Field | 55
  SEC, Week 72, 0.2-0.4/Some Field | 6
  SEC, Week 72, 1-2/Every Field | 5
  SEC, Week 72, 3-5/Every Field | 1
  SEC, Week 72, 6-10/Every Field | 2
  SEC, Week 72, 10-20/Every Field | 1
  SEC, Week 72, 20-30/Every Field | 3
  SEC, Week 84, many/Every Field | 1
  SEC, Week 84, 0-0.1/Some Field | 52
  SEC, Week 84, 0.2-0.4/Some Field | 8
  SEC, Week 84, 1-2/Every Field | 5
  SEC, Week 84, 3-5/Every Field | 4
  SEC, Week 84, 6-10/Every Field | 2
  SEC, Week 96, 0-0.1/Some Field | 56
  SEC, Week 96, 0.2-0.4/Some Field | 4
  SEC, Week 96, 1-2/Every Field | 8
  SEC, Week 96, 3-5/Every Field | 1
  SEC, Week 96, 6-10/Every Field | 2
  SEC, Week 96, 10-20/Every Field | 1
  TEC, Week 60, 0-0.1/Some Field | 3
  TEC, Week 60, 0.2-0.4/Some Field | 1
  TEC, Week 72, 0-0.1/Some Field | 7
  TEC, Week 84, 0-0.1/Some Field | 3
  TEC, Week 96, 0-0.1/Some Field | 5
  UAC, Week 60, 1+ | 1
  UAC, Week 72, 1+ | 1
  UAC, Week 96, 1+ | 2
  WBC, Week 60, 0-0.1/Some Field | 38
  WBC, Week 60, 0.2-0.4/Some Field | 19
  WBC, Week 60, 1-2/Every Field | 12
  WBC, Week 60, 3-5/Every Field | 2
  WBC, Week 60, 6-10/Every Field | 1
  WBC, Week 60, 10-20/Every Field | 1
  WBC, Week 72, 0-0.1/Some Field | 39
  WBC, Week 72, 0.2-0.4/Some Field | 19
  WBC, Week 72, 1-2/Every Field | 7
  WBC, Week 72, 3-5/Every Field | 2
  WBC, Week 72, 6-10/Every Field | 5
  WBC, Week 72, 30-50/Every Field | 1
  WBC, Week 84, many/Every Field | 2
  WBC, Week 84, 0-0.1/Some Field | 47
  WBC, Week 84, 0.2-0.4/Some Field | 12
  WBC, Week 84, 1-2/Every Field | 6
  WBC, Week 84, 10-20/Every Field | 3
  WBC, Week 84, 20-30/Every Field | 1
  WBC, Week 84, 30-50/Every Field | 1
  WBC, Week 96, 0-0.1/Some Field | 41
  WBC, Week 96, 0.2-0.4/Some Field | 18
  WBC, Week 96, 1-2/Every Field | 8
  WBC, Week 96, 6-10/Every Field | 4
  WBC, Week 96, 20-30/Every Field | 1

30. Secondary Outcome: Change From Baseline Values for Beta-2-microglobulin
Description: Urine samples were collected for analysis of urinalysis data for beta-2-microglobulin. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1, Pre-dose) and at Weeks 4, 12, 24, 36, 48, 60, 72, 84 and 96
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Micrograms per liter
Arm/Group | Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 75
Micrograms per liter
  Week 4, n=75 | 206.9 (593.69)
  Week 12, n=74: number analyzed (Participants) | 74
  Week 12, n=74 | 254.6 (891.36)
  Week 24, n=74: number analyzed (Participants) | 74
  Week 24, n=74 | 392.7 (1544.73)
  Week 36, n=73: number analyzed (Participants) | 73
  Week 36, n=73 | 261.1 (715.81)
  Week 48, n=73: number analyzed (Participants) | 73
  Week 48, n=73 | 206.8 (580.77)
  Week 60, n=73: number analyzed (Participants) | 73
  Week 60, n=73 | 309.4 (651.85)
  Week 72, n=73: number analyzed (Participants) | 73
  Week 72, n=73 | 235.7 (542.52)
  Week 84, n=72: number analyzed (Participants) | 72
  Week 84, n=72 | 271.3 (616.86)
  Week 96, n=72: number analyzed (Participants) | 72
  Week 96, n=72 | 196.1 (478.68)

31. Secondary Outcome: Change From Baseline Values for Urine Creatinine Concentration and Urine Phosphate
Description: Urine samples were collected for analysis of urinalysis data for urine creatinine concentration and urine phosphate. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day 1, Pre-dose) and at Weeks 4, 12, 24, 36, 48, 60, 72, 84 and 96
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Milligrams per deciliter
Arm/Group | Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 75
Milligrams per deciliter
  Urine Creatinine, Week 4, n=75 | -5.353 (64.9427)
  Urine Creatinine, Week 12, n=74: number analyzed (Participants) | 74
  Urine Creatinine, Week 12, n=74 | 2.047 (70.1488)
  Urine Creatinine, Week 24, n=74: number analyzed (Participants) | 74
  Urine Creatinine, Week 24, n=74 | 11.715 (78.3996)
  Urine Creatinine, Week 36, n=73: number analyzed (Participants) | 73
  Urine Creatinine, Week 36, n=73 | 15.849 (67.4606)
  Urine Creatinine, Week 48, n=73: number analyzed (Participants) | 73
  Urine Creatinine, Week 48, n=73 | 4.674 (71.2417)
  Urine Creatinine, Week 60, n=73: number analyzed (Participants) | 73
  Urine Creatinine, Week 60, n=73 | 5.567 (58.5998)
  Urine Creatinine, Week 72, n=73: number analyzed (Participants) | 73
  Urine Creatinine, Week 72, n=73 | -1.378 (62.0304)
  Urine Creatinine, Week 84, n=72: number analyzed (Participants) | 72
  Urine Creatinine, Week 84, n=72 | 19.337 (73.2844)
  Urine Creatinine, Week 96, n=72: number analyzed (Participants) | 72
  Urine Creatinine, Week 96, n=72 | 10.346 (69.2155)
  Urine phosphate, Week 4, n=75 | -3.87 (34.392)
  Urine phosphate, Week 12, n=74: number analyzed (Participants) | 74
  Urine phosphate, Week 12, n=74 | -2.08 (35.796)
  Urine phosphate, Week 24, n=74: number analyzed (Participants) | 74
  Urine phosphate, Week 24, n=74 | 2.46 (35.994)
  Urine phosphate, Week 36, n=73: number analyzed (Participants) | 73
  Urine phosphate, Week 36, n=73 | 0.85 (36.016)
  Urine phosphate, Week 48, n=73: number analyzed (Participants) | 73
  Urine phosphate, Week 48, n=73 | 0.68 (36.561)
  Urine phosphate, Week 60, n=73: number analyzed (Participants) | 73
  Urine phosphate, Week 60, n=73 | -0.09 (37.888)
  Urine phosphate, Week 72, n=73: number analyzed (Participants) | 73
  Urine phosphate, Week 72, n=73 | 0.85 (34.012)
  Urine phosphate, Week 84, n=72: number analyzed (Participants) | 72
  Urine phosphate, Week 84, n=72 | 5.21 (34.599)
  Urine phosphate, Week 96, n=72: number analyzed (Participants) | 72
  Urine phosphate, Week 96, n=72 | -0.72 (38.732)

32. Secondary Outcome: Absolute Values for Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Blood pressure of participants were measured at indicated time points in supine position after 5 minutes rest. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose) and at Weeks 4, 12, 24, 36, 48, 60, 72, 84 and 96
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 75
Millimeters of mercury
  SBP, Baseline (Day 1), n=75 | 122.5 (14.15)
  SBP, Week 4, n=75 | 122.9 (12.91)
  SBP, Week 12, n=74: number analyzed (Participants) | 74
  SBP, Week 12, n=74 | 124.9 (16.28)
  SBP, Week 24, n=74: number analyzed (Participants) | 74
  SBP, Week 24, n=74 | 121.9 (12.33)
  SBP, Week 36, n=73: number analyzed (Participants) | 73
  SBP, Week 36, n=73 | 121.5 (14.81)
  SBP, Week 48, n=73: number analyzed (Participants) | 73
  SBP, Week 48, n=73 | 122.5 (14.76)
  SBP, Week 60, n=73: number analyzed (Participants) | 73
  SBP, Week 60, n=73 | 124.7 (14.68)
  SBP, Week 72, n=73: number analyzed (Participants) | 73
  SBP, Week 72, n=73 | 124.2 (15.36)
  SBP, Week 84, n=72: number analyzed (Participants) | 72
  SBP, Week 84, n=72 | 122.1 (12.86)
  SBP, Week 96, n=72: number analyzed (Participants) | 72
  SBP, Week 96, n=72 | 120.8 (16.07)
  DBP, Baseline (Day 1), n=75 | 76.0 (11.76)
  DBP, Week 4, n=75 | 75.2 (11.12)
  DBP, Week 12, n=74: number analyzed (Participants) | 74
  DBP, Week 12, n=74 | 78.1 (10.44)
  DBP, Week 24, n=74: number analyzed (Participants) | 74
  DBP, Week 24, n=74 | 75.6 (10.05)
  DBP, Week 36, n=73: number analyzed (Participants) | 73
  DBP, Week 36, n=73 | 75.3 (10.18)
  DBP, Week 48, n=73: number analyzed (Participants) | 73
  DBP, Week 48, n=73 | 77.8 (11.37)
  DBP, Week 60, n=73: number analyzed (Participants) | 73
  DBP, Week 60, n=73 | 78.0 (11.07)
  DBP, Week 72, n=73: number analyzed (Participants) | 73
  DBP, Week 72, n=73 | 77.5 (10.88)
  DBP, Week 84, n=72: number analyzed (Participants) | 72
  DBP, Week 84, n=72 | 76.3 (10.23)
  DBP, Week 96, n=72: number analyzed (Participants) | 72
  DBP, Week 96, n=72 | 76.1 (10.59)

33. Secondary Outcome: Absolute Values for Heart Rate
Description: Heart rate of participants were measured at indicated time points in supine position after 5 minutes rest. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose) and at Weeks 4, 12, 24, 36, 48, 60, 72, 84 and 96
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 75
Beats per minute
  Baseline (Day 1), n=75 | 74.7 (9.14)
  Week 4, n=75 | 75.8 (10.51)
  Week 12, n=74: number analyzed (Participants) | 74
  Week 12, n=74 | 76.0 (11.05)
  Week 24, n=74: number analyzed (Participants) | 74
  Week 24, n=74 | 74.8 (10.17)
  Week 36, n=73: number analyzed (Participants) | 73
  Week 36, n=73 | 74.3 (9.53)
  Week 48, n=73: number analyzed (Participants) | 73
  Week 48, n=73 | 75.3 (11.32)
  Week 60, n=73: number analyzed (Participants) | 73
  Week 60, n=73 | 75.8 (10.32)
  Week 72, n=73: number analyzed (Participants) | 73
  Week 72, n=73 | 74.9 (11.35)
  Week 84, n=72: number analyzed (Participants) | 72
  Week 84, n=72 | 75.5 (9.96)
  Week 96, n=72: number analyzed (Participants) | 72
  Week 96, n=72 | 73.1 (10.49)

34. Secondary Outcome: Absolute Values for Temperature
Description: Temperature of participants were measured at indicated time points in supine position after 5 minutes rest. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose) and at Weeks 4, 12, 24, 36, 48, 60, 72, 84 and 96
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 75
degrees Celsius
  Baseline (Day 1), n=75 | 36.41 (0.382)
  Week 4, n=75 | 36.43 (0.385)
  Week 12, n=74: number analyzed (Participants) | 74
  Week 12, n=74 | 36.40 (0.448)
  Week 24, n=74: number analyzed (Participants) | 74
  Week 24, n=74 | 36.43 (0.416)
  Week 36, n=73: number analyzed (Participants) | 73
  Week 36, n=73 | 36.45 (0.360)
  Week 48, n=73: number analyzed (Participants) | 73
  Week 48, n=73 | 36.41 (0.414)
  Week 60, n=73: number analyzed (Participants) | 73
  Week 60, n=73 | 36.43 (0.375)
  Week 72, n=73: number analyzed (Participants) | 73
  Week 72, n=73 | 36.42 (0.357)
  Week 84, n=72: number analyzed (Participants) | 72
  Week 84, n=72 | 36.46 (0.349)
  Week 96, n=72: number analyzed (Participants) | 72
  Week 96, n=72 | 36.40 (0.334)

35. Secondary Outcome: Number of Participants With Worst Case Post-Baseline Electrocardiogram (ECG) Values
Description: Twelve-lead ECG was obtained using an ECG machine that automatically calculated the heart rate and measured PR, QRS, QT, and corrected QT (QTc) intervals. Abnormal values with clinically significant and not clinically significant values has been presented. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Time Frame: Up to Week 96
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 75
Participants
  Abnormal-not clinically significant | 20
  Abnormal-clinically significant | 1

36. Secondary Outcome: Change From Baseline Values for Bone Density
Description: Bone densitometry was performed on lumbar spine and femur using dual-energy X-ray absorptiometry (DEXA). Bone density percentage was calculated as bone density observation minus bone density Baseline divided by bone density Baseline. Baseline was considered as Day -1. Change from Baseline is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and at Weeks 24, 48, 72 and 96
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Grams per centimeter^2
Arm/Group | Tenofovir Disoproxil Fumarate
Number analyzed (Participants) | 75
Grams per centimeter^2
  Femur, Week 24, n=0: number analyzed (Participants) | 0
  Femur, Week 48, n=4: number analyzed (Participants) | 4
  Femur, Week 48, n=4 | -0.0125 (0.01654)
  Femur, Week 72, n=0: number analyzed (Participants) | 0
  Femur, Week 96, n=22: number analyzed (Participants) | 22
  Femur, Week 96, n=22 | -0.0205 (0.02765)
  Lumbar vertebra, Week 24, n=1: number analyzed (Participants) | 1
  Lumbar vertebra, Week 24, n=1 | 0.0100 (NA) — NA (Not applicable) indicates standard deviation could not be calculated as a single participant was analyzed.
  Lumbar vertebra, Week 48, n=6: number analyzed (Participants) | 6
  Lumbar vertebra, Week 48, n=6 | -0.0100 (0.04121)
  Lumbar vertebra, Week 72, n=1: number analyzed (Participants) | 1
  Lumbar vertebra, Week 72, n=1 | -0.0620 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed.
  Lumbar vertebra, Week 96, n=72: number analyzed (Participants) | 72
  Lumbar vertebra, Week 96, n=72 | -0.0193 (0.03539)

ADVERSE EVENTS:
Time Frame: SAEs and non-SAEs were collected from the start of the treatment up to Week 96.
Description: SAEs and non-SAEs were collected for Safety Population
Arm/Group | Tenofovir Disoproxil Fumarate
All-Cause Mortality (participants affected / at risk) | 0/75
Serious Adverse Events (participants affected / at risk) | 2/75
Other Adverse Events (participants affected / at risk) | 36/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tenofovir Disoproxil Fumarate (N=75)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Appendicitis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tenofovir Disoproxil Fumarate (N=75)
Beta 2 microglobulin urine increased (Investigations) | 17
Nasopharyngitis (Infections and infestations) | 19
Headache (Nervous system disorders) | 4
Dental caries (Gastrointestinal disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-09-18): https://cdn.clinicaltrials.gov/large-docs/10/NCT03258710/SAP_001.pdf
  • Study Protocol (2018-07-05): https://cdn.clinicaltrials.gov/large-docs/10/NCT03258710/Prot_002.pdf